CLINICAL TRIAL: NCT03921086
Title: Hypertension And Surgery Study 2: A Multicentre, Cross-sectional Quality Improvement Project: Evaluating the Implementation of a Hypertensive Guideline Protocol by Perioperative Clinicians.
Brief Title: Hypertension And Surgery Study: Evaluating the Implementation of a Hypertension Guideline Protocol
Acronym: HASS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Bruce Biccard, Clinical Professor, University of Cape Town
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HASS-2
Record Dates: First submitted 2019-02-20; First posted 2019-04-19 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Hypertension; Metabolic Syndrome; Non-Compliance, Medication
MeSH Terms: conditions — Hypertension; Metabolic Syndrome; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Initiate anti-hypertensive therapy in surgical patients who are identified as hypertensive at the time of their admission. Identify the co-morbidities of these patients (diabetes mellitus, dyslipidemia, renal impairment, obesity and ECG changes)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypertensive patients (Other): Newly diagnosed or poorly controlled hypertensive patients will be initiated on appropriate therapy as per a specific algorithm.
  Interventions: Drug: Antihypertensive medication according to the study's algorithm

INTERVENTIONS:
Drug: Antihypertensive medication according to the study's algorithm — Patients with stage 1 hypertension will receive monotherapy and risks of hypotension are negligible. A single antihypertensive lowers blood pressure (BP) on average by 10/5 mmHg.
  Patients with stage 2 hypertension will be initiated on two medications and this is recommended by all international hypertension guidelines and studies have shown prompt BP control with minimal side effects.
  For borderline patients, the investigators will elect to not treat them for blood pressure ranges of BP: 135-140/85-90 mmHg and give them a letter on discharge to be followed up at their local clinic. The letter will detail that they are potentially hypertensive patients and need to be followed up closely in future.
  Patients with Stage 3 hypertension will be referred to the in-hospital physician as per the algorithm.

SUMMARY:
HASS-2 is a multi-center, cross-sectional quality improvement project: evaluating the implementation of a hypertension guideline protocol by perioperative clinicians, as a model for improving various aspects of public health. The study will also describe the co-morbid risk profile of these newly identified or poorly controlled hypertensive patients. In addition, as a sub-study, these patients will be followed up at monthly intervals for 3 months after discharge, in order to quantify the rates of compliance with their prescribed treatment.

DETAILED DESCRIPTION:
Globally, cardiovascular disease is the leading cause of death. Hypertension is the commonest risk factor underlying cardiovascular disease, and, uncontrolled, is a risk for myocardial infarction, heart failure, stroke and renal disease. Hypertension is common, affecting over 1 billion people worldwide. In modern practice, failure to treat hypertension is regarded as poor medicine, and potentially indefensible.Hypertension remains a global health problem and one that is usually identified and treated in the primary health care setting. However, in South Africa, which is a resource-limited environment, it can burden an already strained primary health care system. The prevalence of hypertension in the adult population of South Africa is approximately 30%. With urbanisation, an ageing population, amongst other developing trends, this number is projected to increase significantly in the future.The perioperative period therefore presents a unique opportunity for clinicians to identify, educate and appropriately initiate or escalate management of these patients, thereby alleviating the burden on the primary health care system.

A short-term quality improvement intervention has the potential to improve quality of care in cardiovascular disease, in a low- to middle-income country like South Africa. This can be done by educating health care providers and implementing a guideline which will lead to improved, standardised and sustained quality of care for patients with hypertension. This will lead to a reduction in blood pressure, and further improve long-term morbidity and mortality of patients, and ultimately reduce the burden on an already strained health care system. Such guidelines could be modified to address other public health care challenges.

Within the African context, South Africans are recognised as being at a significant risk of cardiovascular disease, with the population having the highest prevalence of smoking, dyslipidemia, elevated fasting glucose and abdominal obesity, features of metabolic syndrome.

Metabolic syndrome found in hypertensive patients increases their risk of morbidity and mortality. This, in addition to the added physiological stress of surgery, may dramatically increase cardiovascular risk and complications in this cohort.

Prescribed medications for chronic conditions such as hypertension require a consistent level of patient compliance to the treatment regime. Compliance has been defined as "the extent to which a person's behaviour (in terms of taking medications, following diets or executing lifestyle changes) coincides with medical or health advice". Non-compliance can result in significant implications for not only the patient's health outcomes, but a considerable wastage of resources in an already limited setting. The World Health Organisation has highlighted the considerable economic and health benefits associated with improving compliance with treatments for conditions such as diabetes, hyperlipidaemia and hypertension. Similar to other non-communicable diseases, the ultimate goal of managing hypertension is achieve target control and prevent complications.The secondary aim of the HASS-2 study is to quantify the rates of compliance to antihypertensive medication following discharge from the patient's respective hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Adult (older than 18 years)
* Elective surgery at preoperative in-hospital visit
* All stage 1 and stage 2 hypertensive patients as defined by the South African Hypertension Practice Guideline 2014

Exclusion Criteria:

* Patient refusal
* Day case surgery
* Obstetric and cardiac surgery
* Patients with severe hypertension (>180/110 mmHg) as defined by the South African Hypertension Practice Guideline 2014

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-16 (Actual)

PRIMARY OUTCOMES:
Assessing physician compliance with prescription of in-hospital drugs according to hypertension algorithm | Five day period
  Number of participants who have drugs prescribed in-hospital
Assessing physician compliance with prescription of discharge drugs according to hypertension algorithm | Five day period
  Number of participants who have drugs prescribed at hospital discharge

OTHER OUTCOMES:
Assessing patient compliance with antihypertensive medication dispensing following discharge. | Three and six months following discharge.
  Number of participants who have drugs dispensed following hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Biccard, MD, PhD, Study Director — University of Cape Town
Locations (7):
- South Africa (7):
  - Groote Schuur Hospital, Cape Town, Western Cape
  - Mitchells Plain Hospital, Cape Town, Western Cape
  - Somerset Hospital, Cape Town, Western Cape
  - Victoria Hospital, Cape Town, Western Cape
  - George Hospital, George, Western Cape
  - Paarl Hospital, Paarl, Western Cape
  - Worcester Hospital, Worcester, Western Cape

IPD SHARING:
Plan to Share IPD: No